CLINICAL TRIAL: NCT03056898
Title: Health Professional Dietary Habits and Blood Omega-3 Fatty Acid Concentrations
Status: Completed | Type: Observational
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2016-06-001
Record Dates: First submitted 2017-02-15; First posted 2017-02-17 (Actual); Last update posted 2017-02-20 (Actual); Status verified 2017-02

CONDITIONS: Healthy
Keywords: eicosapentaenoic acid; EPA; docosahexaenoic acid; DHA; omega-3 index

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Health professionals attending the American Association for Family Physicians (AAFP) meeting at the Orlando Convention Center, Sept 21-23, 2016 who visit the DSM Nutritional Products Inc booth will be invited to complete an omega-3 dietary intake survey and have a drop of blood taken by finger stick by a health professional for blood fatty acid analysis. Dried blood samples on filter paper will be sent to an outside laboratory (OmegaQuant LLC) for analysis. Within 2 weeks, participants will receive an Omega-3 Index Test report by email from OmegaQuant LLC. After removing personal information, OmegaQuant LLC will share blood fatty acid and omega-3 dietary intake results with the sponsor.

DETAILED DESCRIPTION:
Omega-3s are important for heart, brain, and joint health. Most Americans have low levels of omega-3s, especially the long-chain fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA), in their blood. The only way to know blood levels of omega-3s is by measurement. The Omega-3 index, a measure of EPA+DHA levels in blood, is determined in a single drop of blood obtained from a finger stick. Blood levels of EPA+DHA can be improved by simple dietary changes.

Twenty-two percent of family physicians report knowing their Omega-3 Index. DSM Nutritional Products Inc will announce the "Know Your O" program at the American Association for Family Physicians (AAFP) meeting at the Orlando Convention Center, Orlando FL, Sept 21-23, 2016 and encourage health professionals to visit the DSM booth (#616) and participate in a dietary survey and have their blood fatty acids measured. After learning more about the study at the DSM Nutritional Products Inc booth, participants will sign an Informed Consent Form, complete an Omega-3 Index Test Request form, and write their name, date of birth and collection date on an OmegaQuant LLC filter paper. Participants will then have a finger stick by a representative from InHouse Physicians, 333 N. Randall Road, Suite 140, St. Charles, IL 60174. Tel (630) 244-0887. Website: www.inhousephysicians.com. The Omega-3 Index Test Request, Informed Consent form and Filter Paper with dried blood sample will be stapled together, packaged with all other samples obtained at that location, and shipped by DSM Nutritional Products Inc to OmegaQuant LLC. Within 2 weeks of receiving the blood sample, OmegaQuant LLC will email the Omega-3 Test results directly to each participant. After removing personal information, OmegaQuant LLC will share blood fatty acid and omega-3 dietary intake results with DSM Nutritional Products Inc for statistical and reporting purposes. DSM Nutritional Products Inc will be unable to link data to any individual. There are no other obligations for participants.

ELIGIBILITY:
Inclusion Criteria:

* Registered member of AAFP with permission to visit exhibitor booths

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health professionals attending the AAFP meeting.
Sampling Method: Non-Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Cross-sectional study of omega-3 fatty acid blood levels | one day
  Single fingerstick to know blood levels of omega-3s

SECONDARY OUTCOMES:
Assessing dietary intake of omega-3 fatty acids | one day
  Self-reported dietary intake

CONTACTS AND LOCATIONS:
Overall Officials: Michael McBurney, PhD, Principal Investigator — DSM Nutritional Products, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harris WS, Von Schacky C. The Omega-3 Index: a new risk factor for death from coronary heart disease? Prev Med. 2004 Jul;39(1):212-20. doi: 10.1016/j.ypmed.2004.02.030. PMID 15208005
- [Derived] Matusheski NV, Marshall K, Hartunian-Sowa S, McBurney MI. US Family Physicians Overestimate Personal omega-3 Fatty Acid Biomarker Status: Associations with Fatty Fish and omega-3 Supplement Intake. Curr Dev Nutr. 2017 Dec 7;2(2):nzx007. doi: 10.3945/cdn.117.002188. eCollection 2018 Feb. PMID 30377677